CLINICAL TRIAL: NCT02532920
Title: The Natural History of Atopic Disease in Thai Children and Association With Atopic March
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Orathai Piboonpocanun, Division of Allergy and Immunology, Department of Pediatrics, Siriraj hospital, Mahidol University
Other Study IDs: 715/2557(EC4)
Record Dates: First submitted 2015-08-20; First posted 2015-08-26 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Atopic Dermatitis
Keywords: Natural history; Atopic dermatitis; Atopic march
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Atopic dermatitis: Atopic dermatitis is diagnosis as Hanifin and Rajka from physician.

SUMMARY:
Atopic dermatitis(AD) is one of manifestation in atopic march. The prevalence of AD is increased. In 1998, the investigators found the prevalence of AD about 15 % in Thailand. AD is diagnosed by clinical as Hanifin and Rajka criteria. There are 3 group of severity defined by SCORAD(Scoring Atopic Dermatitis) : mild (<25), moderate (25-50) and severe (>50). The natural history of AD was mentioned in 3 groups: complete remission, persistent and intermittent. Atopic march is the progression of atopic disease that has atopic dermatitis as the first manifestation then patients will have allergic rhinitis or asthma in the future. The investigators do a retrospective study to understand the natural history of AD as well as it associate with atopic march. That might be a predictive factor of AD and atopic march

DETAILED DESCRIPTION:
Retrospective review from out patient record. Collect the demographic data, onset of atopic march, sensitization of allergen and treatment that given to patients.

For patients who have current follow up at Allergy clinic, the current symptom was collect in that visit.

For patients who didn't have follow up visit, telephone interview was done. If they have symptom, investigators will ask them to come in for investigation and proper treatment.

Patient was recruited in this study with parental permission. The data will collect and use statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AD by physician at birth-15 years old
* Diagnosed by physician by Hanifin and Rajka criteria: itching, dry skin, chronic dermatitis : at face, extensor area (infant), flexor area (children and adult), with or with out history of atopy in family
* Follow at allergy clinic once a year or can ask current symptom via telephone interview.
* Evaluate severity of the disease by SCORAD (Scoring Atopic Dermatitis )

Exclusion Criteria:

* Onset of atopic dermatitis more than 15 years old.
* Other disease: skin, cardiovascular, liver disease, endocrine, neurology, ect
* Not complete data collection in case record form in out patient record.
* Cannot be reach current symptom of patient.

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patient who was diagnosed with atopic dermatitis by physician by searching ICD 10(L20.9, L20.8)
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the natural history of atopic dermatitis in Thai children and the factors that could be associate with the progression of the disease. | Recruited the AD patient who was diagnosed between at birth until 15 years old. The following time at allergy clinic about 4 years in average.
  complete remission (no AD rash and no topical steroid (TS) or topical tacrolimus (TT) use more than one year), persistent (use TS/TT once a month to control AD) and intermittent (other than two groups)

SECONDARY OUTCOMES:
The association of atopic dermatitis and atopic march. | At the first diagnosis of atopic dermatitis until current Allergic visit or telephone interview.The following time at allergy clinic about 4 years in average.

CONTACTS AND LOCATIONS:
Overall Officials: Orathia Piboonpocanun, professor, Study Director — Siriraj Hospital
Locations (1):
- Division of Allergy and Immunology, Department of Pediatrics, Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nicol NH, Boguniewicz M, Strand M, Klinnert MD. Wet wrap therapy in children with moderate to severe atopic dermatitis in a multidisciplinary treatment program. J Allergy Clin Immunol Pract. 2014 Jul-Aug;2(4):400-6. doi: 10.1016/j.jaip.2014.04.009. PMID 25017527
- [Result] Odhiambo JA, Williams HC, Clayton TO, Robertson CF, Asher MI; ISAAC Phase Three Study Group. Global variations in prevalence of eczema symptoms in children from ISAAC Phase Three. J Allergy Clin Immunol. 2009 Dec;124(6):1251-8.e23. doi: 10.1016/j.jaci.2009.10.009. PMID 20004783
- [Result] Chung Y, Kwon JH, Kim J, Han Y, Lee SI, Ahn K. Retrospective analysis of the natural history of atopic dermatitis occurring in the first year of life in Korean children. J Korean Med Sci. 2012 Jul;27(7):723-8. doi: 10.3346/jkms.2012.27.7.723. Epub 2012 Jun 29. PMID 22787365
- [Result] Vichyanond P, Jirapongsananuruk O, Visitsuntorn N, Tuchinda M. Prevalence of asthma, rhinitis and eczema in children from the Bangkok area using the ISAAC (International Study for Asthma and Allergy in Children) questionnaires. J Med Assoc Thai. 1998 Mar;81(3):175-84. PMID 9623008
- [Result] Severity scoring of atopic dermatitis: the SCORAD index. Consensus Report of the European Task Force on Atopic Dermatitis. Dermatology. 1993;186(1):23-31. doi: 10.1159/000247298. PMID 8435513
- [Result] Shaker M. New insights into the allergic march. Curr Opin Pediatr. 2014 Aug;26(4):516-20. doi: 10.1097/MOP.0000000000000120. PMID 24886953
- [Result] Illi S, von Mutius E, Lau S, Nickel R, Gruber C, Niggemann B, Wahn U; Multicenter Allergy Study Group. The natural course of atopic dermatitis from birth to age 7 years and the association with asthma. J Allergy Clin Immunol. 2004 May;113(5):925-31. doi: 10.1016/j.jaci.2004.01.778. PMID 15131576
- [Result] Wisniewski JA, Agrawal R, Minnicozzi S, Xin W, Patrie J, Heymann PW, Workman L, Platts-Mills TA, Song TW, Moloney M, Woodfolk JA. Sensitization to food and inhalant allergens in relation to age and wheeze among children with atopic dermatitis. Clin Exp Allergy. 2013 Oct;43(10):1160-70. doi: 10.1111/cea.12169. PMID 24074334